CLINICAL TRIAL: NCT06348732
Title: Diagnostic and Prognostic Role of Troponin and Brain Natriuretic Peptide in Pediatric Patients With Cardiomyopathy in Correlation to Echocardiography Findings
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan Badawi Hussein, principal investigator, Assiut University
Other Study IDs: biomarkers in cardiomyopathy
Record Dates: First submitted 2024-03-04; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the the role of cardiac biomarkers (troponin and ProBNP) in pediatric Patients with all types of cardiomyopathy in correlation with echocardiography findings .

DETAILED DESCRIPTION:
Cardiomyopathy are structural or functional abnormalities of the myocardium not secondary to congenital, valvular, hypertensive, pulmonary, or coronary heart diseases .

Cardiomyopathy has traditionally been classified into three types based on anatomic and functional features: hypertrophy, dilated, and restrictive. In 1995, two other categories were added by the World Health Organization (WHO), namely, arrhythmical right ventricular cardiomyopathy (dysplasia) (ARVC & ARCD) and unclassified cardiomyopathy .

Over the ensuing years, however, other organizations have proposed or classified cardiomyopathy that emphasize the genetics aspect of the disease.

The original three types of cardiomyopathy are functionally different from one another, and demands of therapy also are different .

In recent years, biomarkers have emerged as important tools for diagnosis, risk stratification and therapeutic decision making in cardiovascular diseases .

Cardiac troponins in particular have become the cornerstone for diagnostic work up of patients with cardiomyopathy. Currently, several promising new biomarkers are under scientific investigation.

Most of these new biomarkers, however, are not yet suitable for clinical application, with exception of B-type natriuretic peptide (BNP) and its N-terminal fragment (NT-ProBNP).

Both markers have proven their diagnostic usefulness in a great number of studies and thus have progressed from bench to clinical application .

This study aims to summarize existing data concerning troponins and NT-ProBNP measurement in pediatric with cardiomyopathy and to outline how these markers can be integrated into clinical routine.

* THE BIOLOGY OF TROPONIN: The 3-unit troponin complex (troponin I, T and C) along with tropomyosin is located on the actin filament and is essential for calcium -mediated regulation of skeletal and cardiac muscle contraction. There is tissue - specific isoforms of troponin I, T and C.

Because the cardiac isoform of troponin C is shared by slow-twitch skeletal muscles, troponin C does not have cardiac specificity and thus is not used in assays of the diagnosis of cardiac injury .

There is one cardiac troponin I (cTn I) isoform in myocardial tissue. This isoform has post-translation tail of 32 amino acids on the N-terminus. This sequence and the 42% and 45% dissimilarity with sequences of other isoforms have made possible the generation of highly specific monoclonal anti-bodies without cross-reactivity with other non-cardiac forms .

Subtypes of troponin (cardiac I and T) are sensitive and specific indicators of heart muscle damage (myocardium).

* B-type natriuretic peptide (BNP) and NT-proBNP in clinical routine: B-type natriuretic peptide, which is also called brain-type natriuretic peptide (BNP), was first described in 1988 after isolation from porcine brain. However, it was soon found to originate mainly from the heart, representing a cardiac hormone.

BNP belongs to the natriuretic peptide family together with other structurally similar peptides, namely atrial natriuretic peptides (ANP), C-type natriuretic peptide (CNP), and Urodilatin .

The natriuretic peptides have in common a characteristic biochemical structure which consists of a 17 amino acid ring and a disulfide bridge between two cysteine molecules. The major source of BNP synthesis and secretion is the ventricular myocardium.

Whereas ANP is stored in granules and can be released immediately after stimulation, only small amounts of BNP are stored in granules and rapid gene expression with de novo synthesis of the peptide is the underlying mechanism of the regulation of BNP secretion .

BNP is synthesized as a prohormone (proBNP) comprising 108 amino acids. Upon release into the circulation it is cleaved in equal proportions into the biologically active 32 amino acid BNP, which represents the C-terminal fragment, and the biologically inactive 76 amino acid N-terminal fragment (NT-proBNP).

Both molecules are constantly released and can be detected in the blood. The main stimulus for increased BNP and NT-proBNP synthesis and secretion is myocardial wall stress .

ELIGIBILITY:
Inclusion Criteria:

Patients more than one month old and younger than 18 years old with any types of cardiomyopathy admitted at Assiut University Children Hospital.

-

Exclusion Criteria:

Patients aged more than 18 years old.

* Patients aged less than one month old .
* Patients with congenital heart diseases .
* Patients with other chronic diseases as : ( chronic kidney diseases , chronic lung diseases, chronic blood diseases and immune deficiency )
* Patients with acute myocarditis secondary to viral infection .

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients more than one month old and younger than 18 years old with any types of cardiomyopathy treated at Assiut University Children Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic and Prognostic Role of Troponin and Pro BNP in Pediatric Patients with Cardiomyopathy in correlation to Echocardiography findings . | one year
  Assess the relation between the outcome of pediatric patients with cardiomyopathy and the serum levels of Troponin and proBNP with echocardiography findings by follow up serum troponin and pro-BNP at months 1, 3, 6 , 9 ,12 in correlation to echocardiography findings and tissue doppler imaging in the assessment of myocardial systolic and diastolic function , All the tissue doppler echocardiographic imaging with systolic and diastolic myocardial velocities will be acquired at the mitral annuli on apical 4-chamber view , in the mitral inflow Doppler velocities examination , peak early diastolic velocity (E) and peak late diastolic velocity (A) will be measured. In themitral annular TDI velocities examination , peak systolic myocardial velocities (S') , peak early diastolic myocardial velocity (E') and peak late diastolic myocardial velocity (A') will be recorded .

REFERENCES:
- [Background] Hamada T, Kubo T, Kitaoka H, Hirota T, Hoshikawa E, Hayato K, Shimizu Y, Okawa M, Yamasaki N, Matsumura Y, Yabe T, Takata J, Doi YL. Clinical features of the dilated phase of hypertrophic cardiomyopathy in comparison with those of dilated cardiomyopathy. Clin Cardiol. 2010 Jul;33(7):E24-8. doi: 10.1002/clc.20533. PMID 20641106
- [Background] Ikeda H, Imaizumi T. [Prognosis of hypertrophic and dilated cardiomyopathy]. Nihon Rinsho. 2000 Jan;58(1):86-92. Japanese. PMID 10885294